CLINICAL TRIAL: NCT03688581
Title: What is the Knowledge and Use of Emergency Contraception for Women Who Are Seeking Abortion in University Hospitals of Strasbourg
Brief Title: What is the Knowledge and Use of Emergency Contraception
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7116
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-09

CONDITIONS: Abortion
Keywords: Abortion; Emergency contraception; Emergency pill; Perception of pregnancy risk; Contraceptive failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to assess the knowledge of women seeking abortion about emergency contraception.

The secondary objectives are to evaluate the use of emergency contraception among women seeking abortion and to identify barriers to the efficacy and use of emergency contraception in these women.

ELIGIBILITY:
Inclusion Criteria:

* women aged over eighteen years old
* the patient agreed that her questionnaire data should be collected and analyzed for this research.
* women who are able to read and write French
* woman seeking an abortion at the Orthogeny Center in University Hospitals of Strasbourg

Exclusion Criteria:

* refusal to participate in the study

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: woman seeking an abortion at the Orthogeny Center in University Hospitals of Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of women's knowledge of contraceptive methods through a questionnaire | 1 hour after consultation for abortion

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologie - CMCO, Strasbourg, France